CLINICAL TRIAL: NCT02178787
Title: UTLight-transcranial Doppler Assessment of Regional Cerebral Autoregulation
Acronym: UTLight
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Ornim Medical Ltd. (Industry)
Responsible Party: Principal Investigator, Vera Novak, Director SAFE laboratory, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2014P000027
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-04

CONDITIONS: Diabetes
Keywords: cerebral blood flow; near infrared spectroscopy; transcranial Doppler; diabetes mellitus; cerebral autoregulation
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 2 diabetes mellitus: Head-up tilt, vasoreactivity, standing up.
- Non-diabetic controls: Head-up tilt, vasoreactivity, standing up.

SUMMARY:
Cerebral autoregulation (CA) is a complex mechanism that serves the essential and vital purpose of controlling cerebral blood flow and metabolism. A stable and optimal brain blood flow is imperative for normal brain function. Diabetes Mellitus (DM ) is associated with microvascular disease that alters CA and also with autonomic failure that may lead to orthostatic hypotension (OH). These conditions may lead to decreased brain blood flow in upright position. This observational study will compare two technologies that evaluate brain blood flow during standing up and other maneuvers in people with and without type 2 diabetes. These technologies are transcranial Doppler and UTLight technology (CerOx). This study will determine the safety and feasibility of CerOx technology for continuous monitoring of cerebral blood flow.

DETAILED DESCRIPTION:
Cerebral autoregulation (CA) is a complex mechanism that serves the essential and vital purpose of controlling cerebral blood flow and metabolism. A stable and optimal brain blood flow is imperative for normal brain function; therefore normal function of CA is crucial for brain health. Diabetes mellitus (DM) is associated with microvascular disease and abnormal autoregulation, which increases risk for stroke and death. Failure of CA has serious consequences across the lifespan and, in terms of prevalence adverse outcomes related to failing CA are most prominent in the elderly with diabetes.

Older diabetic adults often suffer from hypotension or fainting upon standing-up and may have abnormal CA. With abnormal CA, cerebral perfusion and tissue oxygenation declines upon standing up. Abnormalities in perfusion regulation in older people, and particularly those with diabetes may accelerate progression of brain atrophy resulting in cognitive decline, vascular dementia or Alzheimer's disease.

UTLight technology (CerOx), provides a new tool for evaluation of regional blood flow and oxygenation in cortical microvasculature, which is lacking in clinical medicine and patient care. UTLight may become a novel tool that would provide an easy and reliable assessment of regional perfusion and CA in specific cortical areas in health and disease that can be widely implemented in outpatient clinics. This is a pilot, observational feasibility study to compare blood flow measurements using UTLight and TCD.

Aim 1: To assess the safety and feasibility of UTLight for evaluation of regional cerebral blood flow regulation in the anterior circulation ((ACA) and/or middle cerebral artery (MCA) territories) in 20 non-diabetic adults >50 yrs old and 40 age-matched adults with type 2 diabetes.

Aim 2: To compare the profiles of UTLight blood flow (UT_BF), regional oximetry (UT_Ox) and TCD-blood flow velocities (TCD_BFV) in response to: 1) blood pressure changes induced by the postural change from supine to head-up tilt, and from sitting to standing-up; and 2) vasodilatation and vasoconstriction responses induced by hypercapnia and hypocapnia.

The investigators hypothesize that:

1. UT_BF will accurately track TCD_BFV in responses in the anterior circulation (ACA and/or MCA territory) to blood pressure changes, hypercapnia and hypocapnia challenges in healthy older people.
2. UT_BF may be more sensitive to detect abnormalities in regional perfusion in diabetic adults as compared to healthy controls and compared to TCD_BFV.

(UT_Ox) may provide a new indicator to identify older diabetic adults with brain tissue hypoxia during orthostatic challenges that may be at greater risk of brain damage of cognitive decline that will be derived from a change in tissue oxygenation upon standing up that is not routinely evaluated by TCD. Outcomes: Primary outcome is the sensitivity and specificity of UT_BF and TCD_BFV to blood pressure and CO2 challenges, defined as percent change of UT_BF and TCD_BFV in response to hypercapnia and hypocapnia challenges. Secondary outcomes are the differences in cerebral blood flow measured by UT_BF, TCD_BFV between healthy old and diabetic subjects during postural changes. Third outcomes are differences in UT_Ox between healthy old and diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

Diabetes group:

* This group will consist of 40 men and women aged 50-85 years
* diagnosed with type 2 DM and
* treated with oral agents and/or combinations with insulin for at least one year,
* either normotensive [BP <135/85 mm Hg and no medical history of hypertension) or hypertensive [BP >130/85 mm Hg and/or treated for hypertension].

Control group:

* This group will be non-diabetic (normal fasting blood glucose and HbA1c < 6.5%).
* This group will consist of 20 men and women matched with the diabetes group by age ±5 years, and
* subjects will be normotensive [BP <130/85 mm Hg and
* no medical history of hypertension] and
* hypertensive [BP >130/85 mm Hg and/or treated for hypertension].

Exclusion Criteria:

Persons with any one of the following conditions will be excluded:

1. type I diabetes;
2. any unstable or acute medical condition;
3. myocardial infarction or major surgery within 6 months;
4. history of a major stroke;
5. dementia (by history) or inability to follow details of the protocol or MMSE < 20;
6. carotid stenosis > 80% by medical history, Doppler ultrasound, or MR angiography;
7. hemodynamically significant valvular disease;
8. clinically significant arrhythmias;
9. liver or renal failure or transplant;
10. severe hypertension [systolic BP >200 and/or diastolic BP >110 mm Hg or subjects taking ≥3 antihypertensive medications];
11. seizure disorders;
12. malignant tumors;
13. current recreational drug or alcohol abuse;
14. active smoking;
15. morbid obesity (BMI >40).
16. Women in both groups will be required to be postmenopausal.
17. TCD exclusion criteria - poor insonation window and TCD signal;
18. UT_Light exclusion- poor signal.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population sample
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Novak, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventy four consented subjects, thirty type 2 diabetics and thirty non-diabetic controls completed the protocol. Screened participants that did not start the study: eleven were found ineligible after signing informed consent, two withdrew consent, one lost to follow up.
Groups:
- Type 2 Diabetics; Non-diabetic Controls: Head-up tilt, vasoreactivity, sitting to standing-up
Period: Overall Study
Arm/Group | Type 2 Diabetics | Non-diabetic Controls
Started | 35 | 39
Completed | 30 | 30
Not Completed | 5 | 9
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — No TCD window | 3 | 7
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Type 2 Diabetics | Non-diabetic Controls | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7.91) | 66.31 (9.95) | 66.48 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 12 | 18 | 30

OUTCOME MEASURES:

1. Primary Outcome: To Compare Profiles of TCD-blood Flow Velocities (TCD_BFV).
Description: CO2 reactivity will be measured as the slope of regression between TCD_BFV and CO2 changes during baseline, hyperventilation, and CO2 re-breathing.
Time Frame: one year
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Type 2 Diabetics | Non-diabetic Controls
Number analyzed (Participants) | 30 | 30
cm/sec | 28.23 (2.35) | 33.11 (1.54)

2. Secondary Outcome: To Compare Profiles of UTlight Blood Flow (UT_BF) and Regional Oximetry (UT_Ox).
Description: CO2 reactivity will be measured as the slope of regression between UT_BF or UT_Ox and CO2 changes during baseline, hyperventilation, and CO2 re-breathing.
Time Frame: one year
Population: The data analysis has determined that UT_BF and UT_OX signals were not reliable and required further algorithm modification and development during post processing (e.g. raw data signal to noise, signal averaging) that are beyond the scope of the study. Therefore, the results were inconsistent and inconclusive. No results to report.
Arm/Group | Type 2 Diabetes Mellitus | Non-diabetic Controls
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Type 2 Diabetics | Non-diabetic Controls
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Type 2 Diabetics (N=30) | Non-diabetic Controls (N=30)
Headband pressure (Product Issues) | 2 | 1
Lightheadedness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The data analysis has determined that UT_BF signal and UT_OX signals were unreliable and require further development on monitoring algorithm. No results to be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No